CLINICAL TRIAL: NCT03116867
Title: Sonosalpingography in Assessment of Efficacy of Hysteroscopic Tubal Occlusion by Roller Ball Electrode
Brief Title: Sonosalpingography After Hysteroscopic Tubal Occlusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sherif Hanafi Hussain, Assistant Professor, Ain Shams University
Other Study IDs: Ainshams528
Record Dates: First submitted 2017-04-05; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Fallopian Tube Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients receiving hysteroscopic tubal occlusion: This group will have sonosalpingography done for them one month after the tubal occlusion.
  Interventions: Other: sonosalpingography

INTERVENTIONS:
Other: sonosalpingography — transvaginal ultrasound with saline infusion

SUMMARY:
Sonosalpingography is done to assess the efficacy of hysteroscopic tubal occlusion by roller ball electrode.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients with hydrosalpinges requiring in vitro fertilization
* irreversible contraception

Exclusion Criteria:

* Acute pelvic inflammatory disease

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: patients requiring tubal occlusion
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
The presence of fluid in douglas pouch detected by transvaginal ultrasound after saline infusion through the cervix | immediate
  after saline infusion is done, presence of fluid in douglas pouch means that hysteroscopic occlusion of tubes was not successful.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No